CLINICAL TRIAL: NCT03426943
Title: Endotoxins and Cytokines Removal During Continuous Hemofiltration With oXiris™
Acronym: ECRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL17_0014; 2017-A03366-47 (Other: ID-RCB)
Record Dates: First submitted 2018-02-02; First posted 2018-02-08 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2022-10

CONDITIONS: Septic Shock; Peritonitis
MeSH Terms: conditions — Shock, Septic; Peritonitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CVVH using oXiris™ filter (Experimental): Patients included in this arm will have renal replacement therapy by performing Continuous Veno-Venous Hemofiltration (CVVH) using oXiris™ membrane.
  They will also have arterial blood sampling and ultrafiltrate sampling during the CVVH.
  Interventions: Biological: Arterial blood sampling; Biological: Ultrafiltrate sampling; Device: CVVH using oXiris™ filter
- CVVH using PrismafleX HF1400 filter (Active Comparator): Patients included in this arm will have renal replacement therapy by performing CVVH using a standard polysulfone filter (PrismafleX HF1400).
  They will also have arterial blood sampling and ultrafiltrate sampling during the CVVH.
  Interventions: Biological: Arterial blood sampling; Biological: Ultrafiltrate sampling; Device: CVVH using PrismafleX HF1400 filter

INTERVENTIONS:
Biological: Arterial blood sampling — All patients will have arterial blood sampling to assess pre-filter and post-filter plasma endotoxin mass and activity and plasma cytokine levels
Biological: Ultrafiltrate sampling — All patients will have ultrafiltrate sampling to assess cytokine levels
Device: CVVH using oXiris™ filter — Patients included in the experimental arm will have renal replacement therapy by performing CVVH using oXiris™ filter
  Arms: CVVH using oXiris™ filter
Device: CVVH using PrismafleX HF1400 filter — Patients included in the experimental arm will have renal replacement therapy by performing CVVH using PrismafleX HF1400 filter
  Arms: CVVH using PrismafleX HF1400 filter

SUMMARY:
Sepsis is a major cause of death in Intensive Care Units and therefore finding new therapies to improve survival rates and limit morbidity is a major goal. Over the past decades, blood purification has been proposed as an adjuvant therapy for sepsis. The goal of blood purification is to restore the immune homeostasis and efficiency through the removal of bacterial products including endotoxins, broad-spectrum cytokines and other inflammatory mediators. Indeed, the large and overwhelmed release of these mediators in the early phase of sepsis may induce multiple organ failure syndrome. In 2017, different techniques are proposed for blood purification. Among them, the highly adsorptive membrane, oXiris™, seems promising. This membrane can be used in case of Acute Kidney Injury associated with sepsis and exhibits enhanced blood purification capacities. Previous studies on animals have already proven that this membrane can remove broad-spectrum cytokines but also endotoxins from the blood. This ability to remove endotoxins is particularly interesting since endotoxins are believed to be the trigger of the immune cascade at the initiation of sepsis.

The lack of clinical evidence is the main limit to a wider use of this membrane. Therefore, the aim of the present clinical trial is to characterize the blood purification properties of the membrane in a human clinical setting. The oXiris™ membrane is specifically designed to improve the adsorptive capacities of the polyacrylonitrile-based AN69 membrane. Its extremely rich coating of polyethyleneimine (PEI) gives the membrane the ability to bind and remove not only cytokines but also endotoxins due to the positive charges of PEI at the surface of the membrane. The tested hypothesis is that the oXiris™ filter allows for a greater endotoxin and cytokine removal compared to a standard polysulfone ("PrismafleX HF1400") filter in patients with septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 years old,
* "Early" septic shock (in the first 12 hours after Intensive Care Unit (ICU) admission or readmission in the ICU after surgery), with lactatemia > 2 mmol/L and norepinephrine needs > 0.2 µg/kg/min 2 hours after the end of the initial surgery (to ensure that a potential anesthesia effect as disappeared),
* Secondary to a community-acquired or a nosocomial peritonitis (secondary or tertiary but not primary peritonitis),
* AKI KDIGO ≥ stage 2 or another indication for renal replacement therapy, according to the clinician in charge (if baseline creatinine is unknown, KDIGO ≥ stage 2 can be defined by a serum creatinine ≥ 2-fold the normal creatinine for age, gender, and ethnicity).

Exclusion Criteria:

* Inability to obtain informed consent from the patient or next of kin,
* Actual participation in another interventional study,
* Contraindications to citrate,
* Allergy to heparin,
* Pregnant or breastfeeding woman,
* Neutropenia < 0.5 G/L resulting from chemotherapy or other iatrogenic causes
* Patient receiving immunosuppressive therapy, long-term corticosteroids, therapeutic antibodies, chemotherapy in the last 6 months (whatever the dose),
* Patient with innate or acquired immune deficiency (for example severe combined immunodeficiency, HIV or AIDS)
* Onco-hematological disease (lymphoma, leukemia, myeloma) treated within the last 5 years (but inclusion of a patient with solid cancer who did not receive chemotherapy during the past 6 months is possible),
* Patient with expected ICU length of stay < 48 hours,
* Patient for whom a limitation of active care was pronounced at the time of enrollment,
* Patient with no social security insurance, with restricted liberty, or under legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
Interleukin 6 (IL-6) plasmatic concentration | 24 hours after the initiation of CVVH
Endotoxin plasmatic mass concentration | 24 hours after the initiation of CVVH

SECONDARY OUTCOMES:
Pre-filter plasma endotoxin mass | At initiation of CCVH (H0) then 1, 4, 12 and 24 hours after the initiation of CVVH
Pre-filter plasma endotoxin activity | At initiation of CCVH (H0) then 1, 4, 12 and 24 hours after the initiation of CVVH
Post-filter plasma endotoxin mass | 1, 4, 12 and 24 hours after the initiation of CVVH
Post-filter plasma endotoxin activity | 1, 4, 12 and 24 hours after the initiation of CVVH
Pre-filter plasma cytokine level | At initiation of CCVH (H0) then 1, 4, 12 and 24 hours after the initiation of CVVH
Post-filter plasma cytokine level | 1, 4, 12 and 24 hours after the initiation of CVVH
Ultrafiltrate cytokine level | 1, 4, 12 and 24 hours after the initiation of CVVH
Pre-filter plasma lipids level | At initiation of CCVH (H0) then 1, 4, 12 and 24 hours after the initiation of CVVH
Post-filter plasma lipids level | 1, 4, 12 and 24 hours after the initiation of CVVH
Pre-filter plasma Procalcitonin level | At initiation of CCVH (H0) then 1, 4, 12 and 24 hours after the initiation of CVVH
Post-filter plasma Procalcitonin level | 1, 4, 12 and 24 hours after the initiation of CVVH
Pre-filter plasma Phospholipid Transfer Protein level | At initiation of CCVH (H0) then 1, 4, 12 and 24 hours after the initiation of CVVH
Post-filter plasma Phospholipid Transfer Protein level | 1, 4, 12 and 24 hours after the initiation of CVVH
Pre-filter plasma Cholesteryl Ester Transfer Protein level | At initiation of CCVH (H0) then 1, 4, 12 and 24 hours after the initiation of CVVH
Post-filter plasma Cholesteryl Ester Transfer Protein level | 1, 4, 12 and 24 hours after the initiation of CVVH
Pre-filter plasma lipopolysaccharide (LPS) Binding Protein level | At initiation of CCVH (H0) then 1, 4, 12 and 24 hours after the initiation of CVVH
Post-filter plasma LPS-Binding Protein level | 1, 4, 12 and 24 hours after the initiation of CVVH
Norepinephrine requirements | 4, 12 and 24 hours after the initiation of CVVH
Fluids infused | 4, 12 and 24 hours after the initiation of CVVH
Patient survival | At day 7
Patient survival | At day 30
Patient survival | At day 90
Comparison of the results obtained on the above-mentioned parameters, according to the type of bacteria identified from standard care microbiological exams. | At day 7

CONTACTS AND LOCATIONS:
Overall Officials: Thomas RIMMELE, MD, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (8):
- France (8):
  - Hopital Universitaire de Clermont Ferrand, Clermont-Ferrand
  - CHU Francois Mitterrand, Dijon
  - CHU Dijon - Bocage central, Dijon
  - L'Hôpital Nord-Ouest - Villefranche sur Saone, Gleizé
  - Anesthesia and Critical Care Medicine Department - Edouard Herriot Hospital, Lyon
  - Clinique de la Sauvegarde, Lyon
  - Hôpital Pasteur 2 - Hôpital Universitaire de Nice, Nice
  - Hopital Haut Lévèque - CHU Bordeaux, Pessac

REFERENCES:
- [Derived] Tsujimoto Y, Miki S, Shimada H, Tsujimoto H, Yasuda H, Kataoka Y, Fujii T. Non-pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2021 Sep 14;9(9):CD013330. doi: 10.1002/14651858.CD013330.pub2. PMID 34519356